CLINICAL TRIAL: NCT00712478
Title: Observational Study on Efficacy of Intensification of Insulin Therapy to at Least 3 Daily Injections in Type 2 Diabetes
Brief Title: Observational Study Describing Conditions for Intensification of Insulin Therapy in Type 2 Diabetes
Acronym: INTENSE3MIX
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1866
Record Dates: First submitted 2008-06-30; First posted 2008-07-10 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to determine diabetes control improvement, during the third month of follow-up after insulin intensification to at least 3 daily insulin injections, in assessing the proportion of uncontrolled fasting and postprandial glycaemia values recorded on a diary.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients
* Treatment with two insulin daily injections and needing insulin intensification regimen to at least three daily injections
* HbA1c greater than or equal to 8.0%

Exclusion Criteria:

* Patients not performing glycaemia self-measurements
* Secondary diabetes
* Requirement of or use of an insulin pump
* Treatment with corticoids

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 40 years old and more with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluate improvement of diabetes control with fasting glycemia and after diner glycemia measurements | After 3 months

SECONDARY OUTCOMES:
Evaluate improvement of diabetes control with fasting glycemia and after diner glycemia measurements | After first 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Paris La Défense, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com